CLINICAL TRIAL: NCT06103721
Title: Preoperative Dexmedetomidine Nebulization in Blunting Hemodynamic Stress Response to Laryngoscopy
Brief Title: Role of Nebulized Dexmedetomidine in Blunting the Effects of Direct Laryngoscopy and Endotracheal Tube on Heart Rate and Blood Pressure.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Muhammad Haroon Anwar (Other Government)
Collaborators: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Sponsor-Investigator, Muhammad Haroon Anwar, Principal Investigator, Department of Anaesthesia and Critical Care Medicine, Pakistan Institute of Medical Sciences
Organization: Pakistan Institute of Medical Sciences (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: No.F.3-1/2023(ERRB)/Chairman
Record Dates: First submitted 2023-10-16; First posted 2023-10-27 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Hemodynamic Instability
Keywords: Dexmedetomidine; Stress response to laryngoscopy; General Anaesthesia; Direct Laryngoscopy
MeSH Terms: interventions — Dexmedetomidine; Methods; Saline Solution

STUDY DESIGN:
Intervention Model Description: Patients fulfilling the inclusion criteria will be enrolled and divided into two groups through computer generated random numbers. Intervention will be done in the preoperative area under supervision of consultant anesthetist. Afterwards patient will be shifted to operating room, standard ASA monitoring will be attached. General anesthesia will be induced with 1mg of midazolam, 2mg/kg of propofol and 0.5 mg/kg of atracurium. Patient will then be bag mask ventilated for 3 minutes using 100% oxygen at 5 L/min along with Sevoflurane at a MAC (Minimum alveolar concentration) of 1. Vitals will be measured pre-nebulization, pre-induction, and at 1-minute intervals during bag mask ventilation and finally immediately after endotracheal tube placement. Failure to blunt hemodynamic response will be defined as rise in heart rate or blood pressure by more than 20% from pre-induction values immediately after laryngoscopy and endotracheal tube placement which will be managed accordingly.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group Dexmedetomidine (Experimental): This will be the intervention group. Patients entering this group through computer generated random numbers will receive nebulization Dexmedetomidine in the pre-operative area under the supervision of consultant anesthetist.
  Interventions: Drug: Dexmedetomidine Injection [Precedex]
- Group Normal Saline (Placebo Comparator): This will be the placebo or control group. Patients entering this group through computer generated random numbers will receive nebulization with Normal Saline (placebo) in the pre-operative area under the supervision of consultant anesthetist.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Dexmedetomidine Injection [Precedex] — Dexmedetomidine will be diluted in 20 ml of Normal Saline to produce a concentration of 20 mcg/ml. Then it will be taken from the dilution at a dose of 1.0 mcg/kg and that will be added in 2-3 ml of Normal Saline to make it a final volume of 10ml. The resultant mixture will be used to nebulize the patients for 5 minutes, 15 minutes prior to induction of General Anesthesia. Then general anesthesia will be induced with 1mg of Midazolam, 2mg/kg of Propofol, 0.5 mg/kg of Atracurium. Prior to endotracheal tube placement, airway will be managed with bag mask ventilation for 3 minutes. Vitals will be measured pre-nebulization, pre-induction, at 1 minute intervals during bag mask ventilation and immediately after placement of endotracheal tube.
  Other Names: Intervention
  Arms: Group Dexmedetomidine
Drug: Normal Saline — Patients in the placebo group will be nebulized with 10 ml of Normal Saline, 15 minutes prior to induction of general anesthesia. Then general anesthesia will be induced with 1mg of Midazolam, 2mg/kg of Propofol, 0.5 mg/kg of Atracurium. Prior to endotracheal tube placement, airway will be managed with bag mask ventilation for 3 minutes. Vitals will be measured pre-nebulization, pre-induction, at 1 minute intervals during bag mask ventilation and immediately after placement of endotracheal tube.
  Other Names: Placebo
  Arms: Group Normal Saline

SUMMARY:
The goal of this interventional study is to check the effectiveness of nebulized Dexmedetomidine in preventing the rise in blood pressure and heart rate in patients undergoing General Anesthesia. The study will be conducted in patients presenting for elective surgery either healthy or having co-existing medical conditions which affect their daily living to a moderate extent.

These participants will require general anesthesia for their surgical procedure. General Anesthesia will make the patient unconscious, unable to breath and protect his airway.

One way to provide airway and ventilatory support to such patient is by placing endotracheal tube into the patient's windpipe and for that direct laryngoscopy is performed. Direct laryngoscopy is one of the most painful stimulus a person can receive. Therefore like any other thing that causes pain it leads to a rise in blood pressure and heart rate. This can be harmful to the person suffering from cardiac disease.

As a result one must blunt this painful response while providing adequate airway support to the patient needing General Anesthesia. There are number of drugs which can be used for this purpose. They can be given Intravenously or directly into the patient upper airway so that they can make the area numb. One of the drugs which is used for this purpose is Dexmedetomidine.

In this study Dexmedetomidine will be nebulized and directly deliver to the patient's airway just like an asthmatic receives medication from inhaler devices. After giving sufficient time for drug to work, airway will be secured with endotracheal tube using direct laryngoscopy and the degree of rise in Blood Pressure and Heart rate of the patient will be observed. The results will be compared with a control group receiving a substance which looks like a drug but has no effects.

DETAILED DESCRIPTION:
Induction of General Anesthesia results in loss of respiratory drive and protective airway reflexes. This predisposes the person to respiratory failure and aspiration. As a result, airway has to be secured and mechanical ventilation is required. There are numerous ways to secure airway; the most popular being endotracheal tube placement by the help of laryngoscope. Laryngoscopy provides a line of sight from operator's eye to glottis of the patient so that endotracheal tube can be placed. However, laryngoscopy is one of the potent painful stimuli a person can receive. Therefore it results in a number of hemodynamic consequences such as tachycardia and hypertension. This can be problematic for a number of patients such as those with Ischemic Heart Disease, Stenotic Valvular lesions etc.

Blunting this hemodynamic stress response can lead to a number of benefits such as optimal control of hemodynamics. A number of drugs have been used for this purpose such as Lignocaine, Esmolol, Dexmedetomidine, Magnesium Sulphate etc.

Esmolol is a cardio selective beta blocker having a half life of 9 minutes. It blunts the tachycardic and hypertensive response of laryngoscopy. It is given Intravenously.

IV lignocaine given at a dose 1-1.5 mg/kg about 1.5 minutes before intubation can blunt these responses.

Similarly, Dexmedetomidine can be given intravenously to blunt hemodynamic stress response to laryngoscopy. It is an alpha 2 agonist; centrally acting sympatholytic and analgesic agent. Numerous studies and practical experience have shown it be more effective than Beta blockers and Lignocaine. However IV administration of the drug results in hypotension and bradycardia .

If Dexmedetomidine is administered via nebulizer device it can prevent laryngoscopic response as well as its side effects can be minimized.

This study will utilize nebulized Dexmedetomidine to prevent hemodynamic stress response to laryngoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Age: 16 years and above.
* American Society of Anesthesiologists (ASA) class: I, II and III.
* Elective surgeries under General Endotracheal Anesthesia.
* Potentially difficult airway.

Exclusion Criteria:

* Pregnancy
* Body mass index >35 kg/m2
* Known allergy to drugs used in the study
* Liver and renal insufficiency

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Heart Rate | Heart Rate will be assessed pre-nebulization, pre-induction, and at 1 minute intervals during bag mask ventilation, and immediately after endotracheal tube placement.
  Heart Rate is measured as a part of standard ASA monitoring through electronic cardiac monitor showing electrocardiogram as well as heart rate (no. of beats/min).
Blood Pressure | Systolic, Diastolic and Mean arterial blood pressure will be assessed pre-nebulization, pre-induction, and at 1 minute intervals during bag mask ventilation, and immediately after endotracheal tube placement.
  Blood pressure including Systolic, Diastolic and Mean arterial pressure is measured as a part of standard ASA monitoring. This is measured in units of mm of Hg through automated Non-invasive Blood pressure monitoring device.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Haroon Anwar, MBBS, Principal Investigator — Department of Anesthesia and Critical Care, Pakistan Institute of Medical Sciences, Islamabad
Locations (1):
- Deparment of Anesthesia and Critical Care Medicine, Pakistan Institute of Medical Sciences, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Misra S, Behera BK, Mitra JK, Sahoo AK, Jena SS, Srinivasan A. Effect of preoperative dexmedetomidine nebulization on the hemodynamic response to laryngoscopy and intubation: a randomized control trial. Korean J Anesthesiol. 2021 Apr;74(2):150-157. doi: 10.4097/kja.20153. Epub 2020 May 20. PMID 32434291